CLINICAL TRIAL: NCT02137226
Title: Efficacy, Safety and Immunogenicity of BI 695501 Versus Adalimumab in Patients With Active Rheumatoid Arthritis: a Randomized, Double-blind,Parallel Arm, Multiple Dose, Active Comparator Trial
Brief Title: BI 695501 Compared to Adalimumab in Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1297.2; 2012-002945-40 (EudraCT Number)
Record Dates: First submitted 2014-05-12; First posted 2014-05-13 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2017-12

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — BI 695501

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- BI 695501 (Experimental): one injection every 2 weeks for 48 weeks (25 injections in total)
  Interventions: Drug: BI 695501
- US-licensed Humira® (Active Comparator): one injection every 2 weeks for 48 weeks (25 injections in total)
  Interventions: Drug: US-licensed Humira®

INTERVENTIONS:
Drug: BI 695501 — BI 695501, every two weeks for 48 weeks (25 injections in total)
  Arms: BI 695501
Drug: US-licensed Humira® — one injection every 2 weeks for 48 weeks (25 injections in total)
  Arms: US-licensed Humira®

SUMMARY:
Primary Objective:

The primary objective of this trial is to establish an equivalence in efficacy between BI 695501 and US-licensed Humira® in patients with active Rheumatoid arthritis based on a statistical comparison of the proportion of patients meeting American College of Rheumatology 20% (ACR20) response rate at Week 12 and ACR20 response rate at Week 24 between BI 695501 and US-licensed Humira®.

Secondary Objectives:

The secondary objectives of this trial are to compare the efficacy, safety and immunogenicity of BI 695501 and US-licensed Humira® in patients with active RA including those undergoing the transition from US-licensed Humira® to BI 695501 after 24 weeks.

ELIGIBILITY:
Inclusion criteria:

* All patients must sign and date an Informed Consent Form consistent with International Conference on Harmonisation Good Clinical Practice (ICH GCP) guidelines and local legislation prior to participation in the trial (i.e. prior to any trial procedures, which include medication washout and restrictions) and be willing to follow the protocol.
* Male or female participants, between 18 and 80 years of age, who have a diagnosis of moderately to severely active Rheumatoid arthritis for at least 6 months as defined by at least six swollen joints (66 joint count) and at least six tender joints (68 joint count) at Screening and Baseline (Day 1), and either an Erythrocyte sedimentation rate of >28 mm/hour OR a C-reactive protein (CRP) level >1.0 mg/dL (normal: <0.4 mg/dL) at Screening. Patients must currently be receiving methotrexate (MTX) therapy.
* Current treatment for Rheumatoid arthritis on an outpatient basis:

  1. Must be receiving and tolerating oral or parenteral MTX therapy at a dose of 15 to 25 mg per week (dose may be as low as 10 mg per week if the patient is unable to tolerate a higher dose) for at least 12 weeks immediately prior to Day 1. The dose and administration route should remain stable for at least 4 weeks prior to Day 1 until Week 24. After Week 24 the administration route can be changed at the investigator's discretion. Patients receiving a lower dose of MTX (10 to 14 mg/week) should be doing so as a result of a documented history of intolerance to higher doses of MTX.
  2. Patients must be willing to receive oral folic acid (at least 5 mg/week or as per local practice) or folinic acid (at least 1 mg/week or as per local practice) or equivalent during the entire trial (mandatory comedication for MTX treatment).
  3. Disease modifying antirheumatic drug (DMARD) use will be restricted according to guidelines listed in the trial protocol.
  4. If receiving current treatment with oral corticosteroids (other than intra-articular or parenteral), the dose must not exceed 10 mg/day prednisolone or equivalent. During the 4 weeks prior to Baseline (Day 1) the dose must remain stable.
  5. Any concomitant non-steroidal anti-inflammatory drugs (NSAIDs) must be stable for at least 2 weeks prior to Day 1.
  6. Patients may be taking oral hydroxychloroquine provided that the dose is not greater than 400 mg/day or chloroquine provided that the dose is not greater than 250 mg/day. These doses must have been stable for a minimum of 12 weeks prior to Day 1. The hydroxychloroquine or chloroquine treatment will need to be continued at a stable dose with the same formulation until the end of the trial.
* For participants of reproductive potential (males and females), a reliable means of contraception has to be used throughout trial participation(acceptable methods of birth control include for example birth control pills, intrauterine devices [IUDs], surgical sterilization, vasectomized partner and double barrier method.. All patients (males and females of child-bearing potential) must also agree to use an acceptable method of contraception for 6 months following completion or discontinuation from the trial medication.

Exclusion criteria:

* ACR functional Class IV or wheelchair/bed bound.
* Primary or secondary immunodeficiency, including known history of HIV infection, or a positive test at Screening.
* History of Tuberculosis, latent Tuberculosis, or positive purified protein derivative test or interferon gamma-releasing assay .
* Known clinically significant coronary artery disease or significant cardiac arrhythmias or severe congestive heart failure, or interstitial lung disease.
* Previous treatment with >=2 biologic agents.
* Previous treatment with adalimumab or adalimumab biosimilar.
* Current treatment or previous treatment with leflunomide within 8 weeks.
* History of a severe allergic reaction or anaphylactic reaction to a biological agent or history of hypersensitivity to adalimumab or any component of the trial drug.
* History of cancer including solid tumors, hematologic malignancies, and carcinoma in situ.
* Has evidence of positive serology for Hepatitis B virus or Hepatitis C virus
* Receipt of a live/attenuated vaccine within 12 weeks prior to the Screening Visit. Patients who are expecting to receive any live virus or bacterial vaccinations during the trial, or up to 3 months after the last dose of trial drug.
* Any treatment that, in the opinion of the investigator, may place the patient at unacceptable risk during the trial.
* Patients with a significant disease other than Rheumatoid arthritis and/or a significant uncontrolled disease (such as, but not limited to, nervous system, renal, hepatic, endocrine, or gastrointestinal disorders). A significant disease is defined as a disease which, in the opinion of the investigator, may (i) put the patient at risk because of participation in the trial, or (ii) influence the results of the trial, or (iii) cause concern regarding the patient's ability to participate in the trial.
* Premenopausal, sexually active women who are pregnant or nursing, or are of child-bearing potential and not practicing an acceptable method of birth control, or do not plan to continue practicing an acceptable method of birth control throughout the trial.
* History of, or current, inflammatory joint disease other than Rheumatoid arthritis or other systemic autoimmune disorder.
* Diagnosis of juvenile idiopathic arthritis, and/or Rheumatoid arthritis before age 16.
* Any planned surgical procedure within 12 weeks prior to the Screening Visit or for the duration of the trial.
* Known active infection of any kind (excluding fungal infections of nail beds), or any major episode of infection requiring hospitalization or treatment with intravenous anti infectives within 4 weeks of the Screening Visit or completion of oral anti-infectives within 2 weeks of the Screening Visit.
* History of deep space/tissue infection within 52 weeks of the Screening Visit.
* History of serious infection or opportunistic infection in the last 2 years.
* Any neurological, vascular or systemic disorder that might affect any of the efficacy assessments.
* Currently active alcohol or drug abuse or history of alcohol or drug abuse within 2 years of the Screening Visit.
* Treatment with intravenous Gamma Globulin or the Prosorba® Column within 6 months of the Screening Visit.
* Treatment with intravenous, intramuscular, intra-articular and parenteral corticosteroids within 6 weeks prior to Day 1 or throughout the trial.
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 times upper limit of normal.
* Hemoglobin <8.0 g/dL.
* Platelets <100,000/µL.
* Leukocyte count <4000/µL.
* Creatinine clearance <60 mL/min.
* Patients who are currently participating in another clinical trial or who have been participating in another clinical trial with another investigational drug within a minimum of 12 weeks or five half-lives (whichever is longer) of the drug prior to Day 1.
* Patients with a history of any clinically significant adverse reaction to murine or chimeric proteins.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 645 (Actual)
Dates: Start 2015-01-26 (Actual); Primary Completion 2016-03-03 (Actual); Study Completion 2016-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (136):
- United States (61):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Rheumatology Associates, Birmingham, Alabama
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Arizona Arthritis and Rheumatology Research, PLLC, Glendale, Arizona
  - Arizona Arthritis and Rheumatology Research, PLLC, Mesa, Arizona
  - Arizona Arthritis and Rheumatology Research, PLLC, Phoenix, Arizona
  - TriWest Research Associates, LLC, El Cajon, California
  - Advanced Medical Research, LLC, La Palma, California
  - ProHealth Partners, Long Beach, California
  - The Permanente Medical Group, Santa Clara, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - Medvin Clinical Research, Whittier, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Orthopedic Research Institute, Boynton Beach, Florida
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Universal Clinical Research, Coral Gables, Florida
  - Science and Research Institute, Inc., Jupiter, Florida
  - San Marcus Research Clinic, Inc., Miami, Florida
  - L&C Professional Medical Research Institute, Miami, Florida
  - Family Clinical Trials, Incorporated, Pembroke Pines, Florida
  - Physician Research Collaboration, South Miami, Florida
  - West Broward Rheumatology Associates, Incorporated, Tamarac, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - McIlwain Medical Group, PA, Tampa, Florida
  - Lovelace Scientific Resources, Incorporated, Venice, Florida
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - Goldpoint Clinical Research, LLC, Indianapolis, Indiana
  - Heartland Research Associates, LLC, Wichita, Kansas
  - The Arthritis & Diabetes Clinic, Incorporated, Monroe, Louisiana
  - Klein and Associates, M.D., P.A., Cumberland, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Arthritis Education and Treatment Center, Grand Rapids, Michigan
  - North MS Medical Clinics, Incorporated, Tupelo, Mississippi
  - Glacier View Research Institute, Kalispell, Montana
  - Accurate Clinical Research, Inc., Lincoln, Nebraska
  - NJP Clinical Research, Clifton, New Jersey
  - Albuquerque Center For Rheumatology, Albuquerque, New Mexico
  - Anna Imperato, MD PLLC, Manhasset, New York
  - Box Arthritis & Rheumatology of the Carolinas, Charlotte, North Carolina
  - Medication Management, LLC, Greensboro, North Carolina
  - PMG Research of Salisbury, LLC, Salisbury, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - STAT Research, Incorporated, Dayton, Ohio
  - Clinical Research Source, Inc., Perrysburg, Ohio
  - Altoona Center for Clinical Research, P.C., Duncansville, Pennsylvania
  - Mountain View Clinical Research, Greer, South Carolina
  - Center for Inflammatory Disease, Nashville, Tennessee
  - Austin Regional Clinic, Austin, Texas
  - Adriana Pop Moody Clinic PA, Corpus Christi, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Accurate Clinical Management LLC, Houston, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Accurate Clinical Research, Incorporated, Houston, Texas
  - Rheumatology Clinic Of Houston, P.A., Houston, Texas
  - Houston Rheumatology Consultants, PLLC, Houston, Texas
  - Arthritis & Osteoporosis Associates LLP, Lubbock, Texas
  - Accurate Clinical Research, Incorporated, Nassau Bay, Texas
  - Heartland Research Associates, LLC, San Antonio, Texas
  - Danville Orthopedic Clinic, Incorporated, Danville, Virginia
  - Arthritis Northwest, PLLC, Spokane, Washington
- Bulgaria (12):
  - MHAT "Trimontium", OOD, Plovdiv, Plovdiv
  - MHAT "Eurohospital" - Plovdiv, OOD, Plovdiv
  - MHAT - Kaspela, EOOD, Plovdiv
  - Medical Center "Teodora", EOOD, Ruse, Rousse
  - MHAT,Fourth Dept. of Therapeutics & Cardiology, Ruse, Rousse
  - MHAT Shumen AD, Shumen, Shumen
  - MHAT Lyulin, Sofia
  - DCC 17 - Sofia EOOD, Sofia
  - MMA HAT Sofia, Bulgaria, Sofia
  - UMHAT Sv. Ivan Rilski EAD, Sofia
  - DCC 'Chaika', EOOD, Varna, Varna
  - MDHAT 'Dr. Stefan Cherkezov', AD, Veliko Tarnovo
- Chile (6):
  - Corporacion de Beneficencia Osorno, Osorno
  - Quantum Research Santiago, Puerto Varas, Puerto Varas
  - BIOMEDICA, Santiago, Santiago
  - Centro de Estudios Reumatológicos, Santiago
  - Centro Medico Prosalud, Santiago
  - CINVEC - Centro de Investigacion Clinica V Reg.,Vina del Mar, Viña del Mar
- Estonia (2):
  - Pärnu Hospital, Pärnu, Pärnu
  - Medita Kliinik OÜ, Tartu, Tartu
- Germany (4):
  - Rheumazentrum Prof. Dr. G. Neeck, Bad Doberan, Bad Doberan
  - ACURA Kliniken Rheinland-Pfalz AG, Bad Kreuznach, Bad Kreuznach
  - Kerckhoff-Klinik, Bad Nauheim, Bad Nauheim
  - SMO.MD GmbH, Magdeburg, Magdeburg
- Hungary (2):
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klin. Kozpont, Szeged
  - Csolnoky Ferenc Korhaz, Veszprem, Veszprém
- Malaysia (2):
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Hospital Pulau Pinang, Pulau Pinang
- CGM Research Trust, The Princess Margaret Hospital Cantebury, Cantebury, New Zealand
- Poland (12):
  - Gabinet Internistyczno-Reumatologiczny Piotr Adrian Klimiuk, Bialystok
  - Szpital Uniwersytecki nr 2 im.dr J. Biziela, Bydgoszcz
  - Wojewodzki Szpital Zespolony w Elblagu, Elblag
  - Medica Pro Familia Spolka Akcyjna, Oddzial w Gdyni, Gdynia
  - MCBK Iwona Czajkowska Anna Podrazka- Szczepaniak S.C., Grodzisk Mazowiecki
  - Medical Centre Pratia Katowice I, Katowice
  - Medical Centre Pratia Krakow, Krakow
  - Specialist Center ALL-MED, Krakow, Krakow
  - Niepubliczny ZOZ, "Nasz Lekarz", Lekarzy Rodzinnych z, Torun
  - Medical Centre Pratia Warszawa, Warsaw
  - Reumatika, Rheumatology Center, non-public outpatient clinic, Warsaw
  - Wojewodzki Szpital Specjalistyczny we Wroclawiu, Wroclaw
- Russia (8):
  - Kemerovo SMA b/o War Veterans Regional Clinical Hospital, Kemerovo
  - Practicheskaya Meditsina Ltd, Moscow
  - Republic Kareliya Republican Hosp. named after V.A. Baranov, Petrozavodsk
  - Samara Regional Clinical Hospital n.a MI Kalinin, Samara, Samara
  - Reg. Hospital for war veterans, Saratov
  - Stavropol State Medical Academy, Stavropol
  - Emergency Clinical Hospital n. a. N. V. Soloviev, Yaroslavl, Yaroslavl
  - SBHI of Yaroslavl Area "Clinical Hospital #3", Yaroslavl
- Serbia (4):
  - Institute of Rheumatology, Belgrade, Belgrade
  - Institute for Treatment and Rehabilitation, Niska Banja, Niška Banja
  - Clinical Center of Vojvodina, Novi Sad
  - General Hospital "Dr Laza K. Lazarevic" Sabac, Sabac, Šabac
- South Korea (4):
  - Daegu Catholic University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Seoul National University Hospital, Seoul
  - Konkuk University Medical Center, Seoul
- Spain (5):
  - Hospital A Coruña, A Coruña
  - Hospital Universitario de Cruces, Barakaldo
  - Fundación Jiménez Díaz, Madrid
  - Hosp. Nuestra Señora de la Esperanza, Santiago de Compostela, Santiago de Compostela
  - Hospital Clínico de Santiago, Santiago de Compostela
- Thailand (3):
  - Siriraj Hospital, Bangkoknoi
  - Songklanagarind Hospital, Hat Yai
  - Pramongkutklao Hospital, Rajathevee
- Ukraine (10):
  - Ivano-Frankivsk Nat. Medical University, Dept. Endocrinology, Ivano-Frankivsk
  - L.T. Malaya Institute of Therapy AMS of Ukraine, Kharkiv
  - CI of Healthcare Kharkiv CCH #8, Kharkiv, Kharkiv
  - SI NSC M.D. Strazhesko Institute Cardiology of NAMSU, Kyiv, Kyiv
  - SI D.F.Chebotariov Institute of Gerontology of NAMSU, Kyiv, Kyiv
  - Oleksandrivska Clinical Hospital, Kyiv
  - M.V. Sklifosovskyi Poltava RCH, Poltava, Poltava
  - M.I. Pyrogov VRCH, Vinnytsia, Vinnytsia
  - MCIC MC LLC Health Clinic, Vinnytsia, Vinnytsia
  - Zaporizhzhia Regional Clinical Hospital, Zaporizhzhia, Zaporizhzhia

REFERENCES:
- [Derived] Strand V, McCabe D, Bender S. Immunogenicity of adalimumab reference product and adalimumab-adbm in patients with rheumatoid arthritis, Crohn's disease and chronic plaque psoriasis: a pooled analysis of the VOLTAIRE trials. BMJ Open. 2024 Nov 17;14(11):e081687. doi: 10.1136/bmjopen-2023-081687. PMID 39551590
- [Derived] Strand V, Bender S, McCabe D. Effects of Adalimumab-adbm Versus Adalimumab Reference Product on Patient-Reported Outcomes in Rheumatoid Arthritis: Results from VOLTAIRE-RA. Rheumatol Ther. 2024 Oct;11(5):1291-1302. doi: 10.1007/s40744-024-00687-w. Epub 2024 Aug 9. PMID 39120847
- [Derived] Cohen SB, Lee EC. Plain language summary of the VOLTAIRE-RA in patients with moderate-to-severe rheumatoid arthritis. Immunotherapy. 2022 Oct;14(15):1183-1190. doi: 10.2217/imt-2022-0106. Epub 2022 Sep 6. PMID 36065786
- [Derived] Huizinga TWJ, Torii Y, Muniz R. Adalimumab Biosimilars in the Treatment of Rheumatoid Arthritis: A Systematic Review of the Evidence for Biosimilarity. Rheumatol Ther. 2021 Mar;8(1):41-61. doi: 10.1007/s40744-020-00259-8. Epub 2020 Dec 1. PMID 33263165
- [Derived] Kang J, Eudy-Byrne RJ, Mondick J, Knebel W, Jayadeva G, Liesenfeld KH. Population pharmacokinetics of adalimumab biosimilar adalimumab-adbm and reference product in healthy subjects and patients with rheumatoid arthritis to assess pharmacokinetic similarity. Br J Clin Pharmacol. 2020 Nov;86(11):2274-2285. doi: 10.1111/bcp.14330. Epub 2020 Jun 11. PMID 32363771
- [Derived] Cohen SB, Alonso-Ruiz A, Klimiuk PA, Lee EC, Peter N, Sonderegger I, Assudani D. Similar efficacy, safety and immunogenicity of adalimumab biosimilar BI 695501 and Humira reference product in patients with moderately to severely active rheumatoid arthritis: results from the phase III randomised VOLTAIRE-RA equivalence study. Ann Rheum Dis. 2018 Jun;77(6):914-921. doi: 10.1136/annrheumdis-2017-212245. Epub 2018 Mar 7. PMID 29514803

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomized, double-blind, parallel arm, multiple dose, active comparator trial to assess efficacy, safety and immunogenicity of BI 695501 versus adalimumab in patients with active rheumatoid arthritis. Patient received background methotrexate (MTX) treatment.
Pre-assignment Details: One patient was initially treated with Humira and discontinued prior to Week 24. This patient was mistakenly re randomized to BI 695501 but not treated. For safety set this was counted in Humira not re-randomized group (as treated), and for other analysis sets, this patient was counted in the Humira to BI 695501 group (as randomized).
Groups:
- BI 695501: Each patient received 40 milligram (mg)/0.8 millilitre (mL) BI 695501 solution for injection, administered by subcutaneous (SC) injection every 2 weeks up to and including the first 22 weeks of treatment (Period 1).
- US-licensed Humira®: Each patient received 40 mg/0.8 mL US-licenced Humira® solution for injection, administered by SC injection every 2 weeks up to and including the first 22 weeks of treatment (Period 1).
- BI 695501 to BI 695501: Patients initially randomized to BI 695501 in Period 1 and re-randomized to BI 695501 in Period 2. Each patient received 40 mg/0.8 mL BI 695501 solution for injection, administered by SC injection every 2 weeks from Week 24 to Week 48.
- US-licensed Humira® to US-licensed Humira®: Patients initially randomized to US-licensed Humira® in Period 1 and re-randomized to US-licensed Humira® in Period 2. Each patient received 40 mg/0.8 mL US-licenced Humira® solution for injection, administered by SC injection every 2 weeks from Week 24 to Week 48.
- US-licensed Humira® to BI 695501: Patients initially randomized to US-licensed Humira® in Period 1 and re-randomized to BI 695501 in Period 2. Each patient received 40 mg/0.8 mL US-licenced Humira® in period 1 and 40 mg/0.8 mL BI 695501 solution for injection, administered by SC injection every 2 weeks from Week 24 to Week 48.
Period: Period 1 (Initial Randomization)
Arm/Group | BI 695501 | US-licensed Humira® | BI 695501 to BI 695501 | US-licensed Humira® to US-licensed Humira® | US-licensed Humira® to BI 695501
Started | 324 | 321 | 0 | 0 | 0
Completed | 304 (Not completed are discontinued from study) | 305 (Not completed are discontinued from study) | 0 | 0 | 0
Not Completed | 20 | 16 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 5 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 2 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0
Not completed — Other Reason | 1 | 3 | 0 | 0 | 0
Period: Period 2 (Re - Randomization)
Arm/Group | BI 695501 | US-licensed Humira® | BI 695501 to BI 695501 | US-licensed Humira® to US-licensed Humira® | US-licensed Humira® to BI 695501
Started | 0 | 0 | 298 | 148 | 147
Completed | 0 | 0 | 281 (Not completed are discontinued from study) | 140 (Not completed are discontinued from study) | 138 (Not completed are discontinued from study)
Not Completed | 0 | 0 | 17 | 8 | 9
Not completed — Adverse Event | 0 | 0 | 3 | 1 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 8 | 5 | 4
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2 | 0 | 0
Not completed — Other Reason | 0 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF): The SAF contained all patients who received at least one dose of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 695501 | US-licensed Humira® | Total
Number analyzed (Participants) | 324 | 321 | 645
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.7 (12.04) | 53.6 (11.32) | 53.6 (11.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 267 | 269 | 536
  Male | 57 | 52 | 109

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients Meeting the American College of Rheumatology 20% (ACR20) Response Criteria at Week 12
Description: The proportion of patients meeting the ACR20 response criteria was assessed. A patient had an ACR20 response if all of the following occurred: A ≥ 20 % improvement in the swollen joint count (66 joints), A ≥ 20 % improvement in the tender joint count (68 joints), A ≥ 20 % improvement in at least three of the following assessments: Patient's assessment of pain, Patient's global assessment of disease activity (equivalent to the General Health component of the Disease Activity Score (DAS)), Physician's global assessment of disease activity, Patient's assessment of physical function, as measured by the Health Assessment Questionnaire - Disability Index (HAQ-DI) Acute phase reactant (C-reactive protein (CRP)).The Full Analysis Set contained all enrolled patients who were randomized to trial drug and who received at least one dose of trial drug and had all efficacy measures relevant for the co-primary efficacy endpoints measured at baseline and at least once post- baseline.
Time Frame: Week 12
Population: Full Analysis Set. Patients who discontinued treatment prior to the time-point had their binary response imputed as non-responder, a method commonly known as non-responder imputation. For truly missing data at the component level, multiple imputation was used.
Measure: Number; unit: Percentage of Patients
Arm/Group | BI 695501 | US-licensed Humira®
Number analyzed (Participants) | 321 | 318
Percentage of Patients | 67.0 | 61.1
Statistical Analysis 1: Comparison: BI 695501 vs US-licensed Humira®; The week 12 confidence interval for the estimated difference in proportion is produced using the cumulative distribution function method of Reeve; Test type: Non-Inferiority or Equivalence — The 90% Confidence Interval (CI) for ACR20 at Week 12, rounded to 1 decimal place, had to be entirely contained in the predefined equivalence region [-12.0%, 15.0%]; Regression, Logistic; Difference in proportions = 5.9, 90% CI 2-sided [-0.9 to 12.7] — Results from logistic regression model adjusted for treatment, prior exposure to a biologic agent (yes / no), Baseline DAS28 (ESR). Difference in ACR20 Response Rate (BI695501 - Humira, %) is presented

2. Secondary Outcome: Change From Baseline in Disease Activity Score 28 (DAS28) (Erythrocyte Sedimentation Rate [ESR]) at Week 12 and Week 24
Description: The DAS28 (ESR) score was derived using the following formulae:
  DAS28 (ESR) = 0.56*√(TJC28) + 0.28*√(SJC28) + 0.014*(GH) + 0.7*ln(ESR)
  Where:
  * TJC28 = 28 joint count for tenderness
  * SJC28 = 28 joint count for swelling
  * Ln (ESR) = natural logarithm of ESR
  * GH = General Health component of the DAS (patient's global assessment of disease activity). DAS28 values range from 2.0 to 10.0 while higher values mean a higher disease activity. Actual number of patient analysed (N) is mean number of subjects in the analysis set with DAS28(ESR) results computable across the multiply imputed data sets. It is 319.6, 317.1 for week 12 and 313.9, 315.1 for week 24 for BI 695501 and US-licensed Humira® respectively.
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | BI 695501 | US-licensed Humira®
Number analyzed (Participants) | 321 | 318
Units on a scale
  Week 12 | -2.1 [-2.28 to -2.01] | -2.0 [-2.18 to -1.91]
  Week 24 | -2.4 [-2.51 to -2.21] | -2.4 [-2.54 to -2.24]
Statistical Analysis 1: Comparison: BI 695501 vs US-licensed Humira®; Results based on DAS28 (ESR) mean changes from Baseline after 12 weeks of treatment = overall mean + treatment group + Baseline DAS28 (ESR) + prior exposure to a biologic agent + random error; Test type: Non-Inferiority or Equivalence — Equivalence margin is not applicable; ANCOVA; Mean Difference (Final Values) = -0.1, 90% CI 2-sided [-0.25 to 0.05] — Difference in least square means of BI 695501 - Humira is presented
Statistical Analysis 2: Comparison: BI 695501 vs US-licensed Humira®; Results based on DAS28 (ESR) mean changes from Baseline after 24 weeks of treatment = overall mean + treatment group + Baseline DAS28 (ESR) + prior exposure to a biologic agent + random error; Test type: Non-Inferiority or Equivalence — Equivalence margin is not applicable; ANCOVA; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.17 to 0.23] — Difference in least square means of BI 695501 - Humira is presented

3. Secondary Outcome: The Percentage of Patients With Investigator-assessed Drug-related Adverse Events (AEs) During the Treatment Phase
Description: The analysis of AEs was based on the concept of treatment-emergent AEs (TEAEs). Thus, all AEs with an onset after the first dose of trial drug up to a period of ten weeks after the last dose of trial drug were assigned to the current treatment for evaluation. Investigator-assessed drug related AEs were AEs with a relationship to drug ticked "yes" according to the Investigator. Overall results are presented from Day 1 up to Week 58 and are based on the initial randomization groups. The comparison therefore focuses on patients who received BI 695501 continuously versus patients who received Humira® continuously for the long term assessment of safety. One patient was initially treated with Humira and discontinued prior to Week 24. This patient was mistakenly re randomized to BI 695501 but not treated. For safety this was counted in Humira not re-randomized group (as treated), and for other analysis sets, this patient was counted in the Humira to BI 695501 group (as randomized).
Time Frame: From the first drug administration until 10 weeks after the last drug administration, up to 58 weeks
Population: The Safety Analysis Set contained all patients who received at least one dose of trial drug.
Measure: Number; unit: Percentage of Patients
Groups:
- BI 695501 Continuously: BI 695501 continuously comprised all patients randomized to BI 695501 in Period 1 and re-randomized to BI 695501 in Period 2 (or not re randomized at Week 24). This group represents all patients who were to receive BI 695501 from Day 1 to Week 48. Each patient received 40 mg/0.8 mL BI 695501 solution for injection, administered by SC injection every 2 weeks.
- US-licensed Humira® Continuously: Humira® US continuously comprised all patients randomized to US-licensed Humira® in Period 1 and re-randomized to US-licensed Humira® in Period 2 or not re randomized at Week 24 (e.g. patients who discontinued treatment prior to Week 24). This group represents all patients who were to receive US-licensed Humira® from Day 1 to Week 48. Each patient received 40 mg/0.8 mL US-licensed Humira® solution for injection, administered by SC injection every 2 weeks.
Arm/Group | BI 695501 Continuously | US-licensed Humira® Continuously
Number analyzed (Participants) | 324 | 175
Percentage of Patients | 19.1 | 22.9

4. Primary Outcome: The Proportion of Patients Meeting ACR20 Response Criteria at Week 24
Description: ACR20 at Week 12 and Week 24 are standard outcome criteria that are widely accepted for regulatory purposes to demonstrate efficacy in treating the signs and symptoms of Rheumatoid arthritis (RA). The proportion of patients meeting the ACR20 response criteria was assessed at Week 12 and Week 24 to provide a robust comparison with US-licensed Humira® data. A patient had an ACR20 response if all of the following occurred: A ≥ 20 % improvement in the swollen joint count (66 joints), A ≥ 20 % improvement in the tender joint count (68 joints), A ≥ 20 % improvement in at least three of the following assessments: Patient's assessment of pain, Patient's global assessment of disease activity (equivalent to the General Health component of the Disease Activity Score ([DAS]), Physician's global assessment of disease activity, Patient's assessment of physical function, as measured by the Health Assessment Questionnaire - Disability Index (HAQ-DI) Acute phase reactant (C-reactive protein [CRP]).
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | BI 695501 | US-licensed Humira®
Number analyzed (Participants) | 321 | 318
Percentage of Patients | 69.0 | 64.5
Statistical Analysis 1: Comparison: BI 695501 vs US-licensed Humira®; The week 24 confidence interval for the estimated difference in proportion is produced using the cumulative distribution function method of Reeve; Test type: Non-Inferiority or Equivalence — The 95% Confidence Interval (CI) for ACR20 at Week 24, rounded to 1 decimal place, had to be entirely contained in the predefined equivalence region [-15.0%;+15.0%]; Regression, Logistic; Difference in proportions = 4.5, 95% CI 2-sided [-3.4 to 12.5] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From the first drug administration until 10 weeks after the last drug administration, up to 58 weeks
Description: Treatment-emergent adverse events are defined as adverse events that started or worsened on or after the first dose of study medication and prior to the last date of study medication plus 10 weeks (70 days) inclusive. Data is reported from Day 1 to the end of Period 2 (Week 58).
Arm/Group | BI 695501 Continuously | US-licensed Humira® Continuously
Serious Adverse Events (participants affected / at risk) | 18/324 | 17/174
Other Adverse Events (participants affected / at risk) | 35/324 | 24/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695501 Continuously (N=324) | US-licensed Humira® Continuously (N=174)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Hypertensive cardiomyopathy (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Macular degeneration (Eye disorders) | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 3
Pyelonephritis acute (Infections and infestations) | 0 | 2
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint destruction (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695501 Continuously (N=324) | US-licensed Humira® Continuously (N=174)
Nasopharyngitis (Infections and infestations) | 19 | 17
Upper respiratory tract infection (Infections and infestations) | 17 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.